CLINICAL TRIAL: NCT04402697
Title: Study of the Usefulness of Blood Cells for the Analysis of Metabolic Recovery After Weight Loss (METAHEALTH-TEST)
Brief Title: Analysis of Metabolic State in Normal-weight and Overweight-obese After Lifestyle Improvement and/or Weight Loss
Acronym: METAHEALTH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Balearic Islands (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: nºIB 3216/16 PI
Record Dates: First submitted 2020-05-13; First posted 2020-05-27 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Overweight and Obesity
Keywords: Overweight; Obesity; Blood cells; Metabolic health; Weight loss
MeSH Terms: conditions — Overweight; Obesity; Weight Loss | interventions — Diet

STUDY DESIGN:
Intervention Model Description: Volunteers are assigned to three groups for the duration of the study:
  1. Normal-weight
  2. Overweight-Obese
  3. Metabolically obese normal-weight
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Normal-weight (NW) (No Intervention): Individuals with BMI<25 kg/m2
- Overweight-Obese (OW-OB) (Experimental): Individuals with BMI>25 kg/m2, submitted to a nutritional intervention (hypocaloric balanced diet) during 6 months and prescription of physical activity to achieve weigh loss
  Interventions: Other: Dietary and physical activity intervention
- Metabolically obese normal-weight (MONW) (Experimental): Individuals with BMI<25 kg/m2, with metabolic alterations related to obesity (hypertriglyceridemia, hypercholesterolemia, hyperglycaemia, hypertension or high waist-hip ratio), submitted to an intervention to improve dietary habits and physical activity in order to achieve a better body composition and metabolic health. Mediterranean diet will be and aerobic and strength exercises will be advised to these individuals.
  Interventions: Other: Dietary and physical activity intervention

INTERVENTIONS:
Other: Dietary and physical activity intervention — OW-OB group: 6-month program of weight loss consisting in a low-calorie food plan (30% reduction in the individual energy requirements) with dietary sessions and exercise counselling.
  MONW group: 6-month program to improve eating habits (Mediterranean diet) with dietary sessions and exercise counselling.
  Arms: Metabolically obese normal-weight (MONW); Overweight-Obese (OW-OB)

SUMMARY:
The aim of this study is to design and validate a test, METAHEALTH-TEST, based in gene expression analysis in blood cells, to quickly and easily analyse metabolic health. This test will be used to analyse metabolic improvement in overweight/obese individuals and in metabolically obese normal-weight (MONW) individuals after undergoing a weight loss intervention and/or an intervention for improvement in eating habits and lifestyle.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-45 years
* Participants with no chronic disease (excluding those related to overweight/obesity)

Exclusion Criteria:

* Minors or older than 45 years
* Presence of a metabolic illness
* Intake of regular medication or drugs
* Precedents of alcohol or drug consumption
* Physic of psychic disability

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2016-05-25 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Number of individuals responding to fasting assessed by changes in gene expression profile of blood cells | Baseline point (all groups)
  The effect of fasting on gene expression profile of blood cells will be analyzed by real-time RT-qPCR and microarray
Number of individuals responding to fasting assessed by changes in gene expression profile of blood cells | 3 months (OW-OB and MONW groups)
  The effect of fasting on gene expression profile of blood cells will be analyzed by real-time RT-qPCR and microarray
Number of individuals responding to fasting assessed by changes in gene expression profile of blood cells | 6 months (OW-OB and MONW groups)
  The effect of fasting on gene expression profile of blood cells will be analyzed by real-time RT-qPCR and microarray
Weight | Baseline point (all groups)
  Weight (kg)
Weight | 3 months (OW-OB and MONW groups)
  Weight (kg)
Weight | 6 months (OW-OB and MONW groups)
  Weight (kg)
Body Mass Index (BMI) | Baseline point (all groups)
  Weight and height will be combined to report BMI in kg/m^2).
Body Mass Index (BMI) | 3 months (OW-OB and MONW groups)
  Weight and height will be combined to report BMI in kg/m^2).
Body Mass Index (BMI) | 6 months (OW-OB and MONW groups)
  Weight and height will be combined to report BMI in kg/m^2).
Body composition | Baseline point (all groups)
  Body composition (fat mass in kg) measured using a DXA scanner
Body composition | 3 months (OW-OB and MONW groups)
  Body composition (fat mass in kg) measured using a DXA scanner
Body composition | 6 months (OW-OB and MONW groups)
  Body composition (fat mass in kg) measured using a DXA scanner
Circulating glucose, triglycerides (TG), total cholesterol, high-density lipoprotein cholesterol (HDL-C), low-density lipoprotein cholesterol (LDL-C), and C-reactive protein (CRP) | Baseline point (all groups)
  Circulating parameters measured in mg/dL
Circulating glucose, triglycerides (TG), total cholesterol, high-density lipoprotein cholesterol (HDL-C), low-density lipoprotein cholesterol (LDL-C), and C-reactive protein (CRP) | 3 months (OW-OB and MONW groups)
  Circulating parameters measured in mg/dL
Circulating glucose, triglycerides (TG), total cholesterol, high-density lipoprotein cholesterol (HDL-C), low-density lipoprotein cholesterol (LDL-C), and C-reactive protein (CRP) | 6 months (OW-OB and MONW groups)
  Circulating parameters measured in mg/dL
Circulating gamma-glutamyl transpeptidase (GGT) | Baseline point (all groups)
  GGT measured in U/L
Circulating gamma-glutamyl transpeptidase (GGT) | 3 months (OW-OB and MONW groups)
  GGT measured in U/L
Circulating gamma-glutamyl transpeptidase (GGT) | 6 months (OW-OB and MONW groups)
  GGT measured in U/L

SECONDARY OUTCOMES:
Height | Baseline point (all groups)
  Height (m)
Height | 3 months (OW-OB and MONW groups)
  Height (m)
Height | 6 months (OW-OB and MONW groups)
  Height (m)
Waist-hip ratio | Baseline point (all groups)
  Waist-hip ratio
Waist-hip ratio | 3 months (OW-OB and MONW groups)
  Waist-hip ratio
Waist-hip ratio | 6 months (OW-OB and MONW groups)
  Waist-hip ratio
Blood pressure | Baseline point (all groups)
  Blood pressure (mm Hg)
Blood pressure | 3 months (OW-OB and MONW groups)
  Blood pressure (mm Hg)
Blood pressure | 6 months (OW-OB and MONW groups)
  Blood pressure (mm Hg)

CONTACTS AND LOCATIONS:
Locations (1):
- University of the Balearic Islands, Palma de Mallorca, Balearic Islands, Spain

IPD SHARING:
Plan to Share IPD: Undecided
IPD will be shared in due time if considered relevant for other research. With our current objectives, it is not considered necessary.

REFERENCES:
- [Derived] Costa A, Konieczna J, Reynes B, Martin M, Fiol M, Palou A, Romaguera D, Oliver P. CUN-BAE Index as a Screening Tool to Identify Increased Metabolic Risk in Apparently Healthy Normal-Weight Adults and Those with Obesity. J Nutr. 2021 Aug 7;151(8):2215-2225. doi: 10.1093/jn/nxab117. PMID 33978191